CLINICAL TRIAL: NCT06415903
Title: A Phase I Study to Evaluate the Safety and Tolerance of TQB3117 Tablets in Patients With Advanced Malignant Cancer
Brief Title: A Clinical Trial of TQB3117 Tablets in Patients With Advanced Malignant Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3117-I-01
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-01

CONDITIONS: Advanced Malignant Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3117 tablets (Experimental): TQB3117 tables is administered as a single dose or multiple dose, ranging from 20 to 180 mg once daily. Oral administration on fast condition, with each cycle lasting 21 days.
  Interventions: Drug: TQB3117 tablets

INTERVENTIONS:
Drug: TQB3117 tablets — TQB3117 is a protein inhibitor.

SUMMARY:
The study is divided into two phases: dose escalation and dose extension. The dosing regimens include a single-dose study and a multiple-dose study. It adopts a single-center, open-label, non-randomized, single-arm clinical trial design, where patients with advanced malignant cancer are selected to orally take TQB3117 tablets. The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of TQB3117 tablets in patients.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study;
* Age: 18 to 75 years old; an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Has at least one assessable lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria;
* The main organs function well;
* Female patient had no plans to become pregnant and voluntarily took effective contraceptive measures from agree with the study to at least 6 months after the last dose of study drug.

Exclusion Criteria:

* There were other malignant tumors in 3 years;
* Has multiple factors affecting oral medication;
* Unalleviated toxicity ≥ grade 1 above CTCAE v5.0 due to any previous therapy, excluding hair loss;
* Major surgical treatment, open biopsy and obvious traumatic injury were performed within 28 days before the study, or have not fully recovered from previous surgery, or are expected to require major surgical surgery during the study period;
* Arteriovenous thrombotic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism;
* Have a history of psychotropic drug abuse and can not quit or have mental disorders;
* Subjects with any severe and / or uncontrolled disease included: active hepatitis, have a history of immunodeficiency;
* Has known symptomatic central nervous system metastases and/or cancerous meningitis;
* Thoracic/abdominal/pericardial effusion with clinical symptoms or requiring repeated drainage, or drainage for the purpose of receiving treatment within one month after receiving the investigational drug for the first time;
* Has participated in other clinical trials within 4 weeks before first dose;
* According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (each cycle is 21 days)
  DLT refers to occurrence of drug-related adverse events within the first treatment cycle after subjects receive single-dose or multiple-dose treatment, as defined by the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 toxicity assessment criteria.
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 21 days)
  MTD is defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Recommended Phase II Dose (RP2D) | Baseline up to 24 months
  DLT describes side effects of a drug or other treatment that are serious enough to evaluate RP2D of TQB3117 tablets in adult patients with advanced malignant cancer.

SECONDARY OUTCOMES:
Adverse events (AE) | 30 days after the last administration
  The occurrence of all adverse events (AE).
Serious adverse events (SAE) | 30 days after the last administration
  The occurrence of all serious adverse events (SAE).
Time to reach maximum plasma concentration (Tmax) | Day 1 of single dose: pre-dose, at 0.5,1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours after-dose. Days 7,14 and 21 of cycle1: pre-dose. Day 21of cycle1: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose.
  To characterize the pharmacokinetics of TQB3117 by assessment of time to reach maximum plasma concentration after single and multiple dosing.
Peak concentration (Cmax) | Day 1 of single dose: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours after-dose. Days 7,14 and 21 of cycle1: pre-dose. Day 21 of cycle 1: at 0.5,1, 2, 3, 4, 6, 8, 12, 24 hours after-dose.
  The maximum observed plasma concentration of study drug.
Half-life (t1/2) | Day 1 of single dose: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours after-dose. Days 7, 14 and 21 of cycle 1: pre-dose. Day 21 of cycle 1: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose.
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Area under the concentration-time curve (AUC [0-infinity] | Day 1 of single dose: pre-dose, at 0.5,1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours after-dose. Days 7, 14 and 21 of cycle 1: pre-dose, Day 21 of cycle 1: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose.
  To characterize the pharmacokinetics of TQB3117 by assessment of area under the plasma concentration time curve from 0 extrapolated to infinity.
Area under the concentration-time curve (AUC [0-t] | Day 1 of single dose: pre-dose, at 0.5,1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours after-dose. Days 7, 14 and 21 of cycle 1: pre-dose. Day 21 of cycle 1: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose.
  To characterize the pharmacokinetics of TQB3117 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Apparent clearance (CL/F) | Day 1 of single dose: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours after-dose. Days 7, 14 and 21 of cycle 1: pre-dose. Day 21 of cycle 1: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose.
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Apparent volume of distribution (Vd/F) | Day 1 of single dose: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours after-dose. Days 7, 14 and 21 of cycle 1: pre-dose. Day 21 of cycle 1: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose.
  Apparent volume of distribution of the TQB3117 in plasma.
Objective Response Rate (ORR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100weeks
  The percentage of complete response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China